CLINICAL TRIAL: NCT02687269
Title: Ranolazine Myocardial Protection in Complete Coronary Artery Bypass Grafting: A Randomized-controlled Trial
Brief Title: Ranolazine a Potential New Therapeutic Application
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to produce placebo tablets similar to the drug tested
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Temistocle Taccheri, MD, Resident in Anesthesia and Intensive Care Department, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RAN
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Stunning
Keywords: myocardial protection; coronary artery bypass grafting
MeSH Terms: conditions — Myocardial Stunning | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranolazine (Experimental): The patients undergoing elective and complete CABG revascularization performed by the same surgeon, will be randomized in two different groups to receive, in the three days before surgery, Ranolazine at a dose of 375 mg twice daily.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): The patients undergoing elective and complete CABG revascularization performed by the same surgeon, will be randomized in two different groups to receive, in the three days before surgery, placebo twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Patients in this arm receive Ranolazine at a dose of 375 mg twice daily in the three days before surgery
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Patients receive Placebo twice daily in the three days before surgery
  Arms: Placebo

SUMMARY:
Despite surgical and medical innovation have reduced mortality rates in cardiac surgery, the disease severity and operative procedural complexity have increased and morbidity rate is still high. Ischemia-reperfusion (I/R) injury, redefined in cardiac surgery "post-cardioplegic injury" (2) as a whole of ischemia-reperfusion, cardiopulmonary bypass and surgical trauma, has been recognized as a significant contributor to mortality and morbidity. I/R injury is classified as reversible or irreversible. Reversible injury includes arrhythmias, edema, vascular dysfunction and contractile stunning expressed as low output syndrome without cell death and without apparent signs of infarction or other serum injury markers. Irreversible reperfusion injury includes apoptosis and necrosis. I/R injury is a complex process associated with increase of radical, oxidant and cytokines production, complement and neutrophil activation and endothelial activation leading to microvascular dysfunction and deterioration of coronary flow reserve. In the hypoxic heart increase anaerobic lactate production, K+ efflux and membrane depolarization. The intracellular Na+ concentration rises as a consequence of slow Na+ channels inactivation and the induction of voltage-gated Na+ channel late current component (late INA). Intracellular Na++ accumulation enhanced activity of reversed-mode Na+-Ca++ exchanger causing intracellular Ca++ overload and ventricular dysfunction. Therefore inhibition of late INA has been shown to be cardioprotective. Ranolazine, an FDA-approval antianginal and anti-ischemic agent, high selective blocker of late INA, inhibits the late sodium current in myocardial ischemia, decreases Na+ and Ca2+ overload and improves left ventricular function in experimental animal models. For this reason it was also adjuncted to cardioplegia improving diastolic function in isolate Langerdoff-perfused rat hearts. The authors test the hypothesis that ranolazine improve myocardical protection in patients undergoing coronary artery surgery with cardiopulmonary by-pass (CPB).

DETAILED DESCRIPTION:
We aim to perform a prospective, single-center, investigator-initiated, randomized (1:1), blinded, placebo-controlled study. The patients undergoing elective and complete CABG revascularization performed by the same surgeon, will be randomized in two different groups to receive, in the three days before surgery, Ranolazine at a dose of 375 mg twice daily or placebo. After the enrollement in the research according the inclusion and exclusion criteria, the randomization list will be computer-generated. The study participants, the reserchers responsible for data reporting and analysis and the ecocardiographers will be blinded to the treatment that each patient will receive. In a previous phase all data for the recruitment will be considered and registered before surgery: basic clinical parameters (age, gender, height, weight, body surface, systolic blood pressure and diastolic blood pressure, mean heart rate); medical history (diabetes mellitus type I or II, smoking status, chronic obstructive pulmonary desease, systemic arterial hypertension, dyslipidemia, family history of cardiovascular events, angina, percutaneous coronary interventions (PCI), acute myocardial infarction (AMI), previous cardiac surgery, chronic peripheral arterial disease, cerebral ischemia, bleeding and chronic renal failure); basic hematologic parameters (creatinine, glucose, hemoglobin, hematocrit, white blood cell counts and equation, platelets number, aPTT, INR); baseline transthoracic echocardiographic (TTE) parameters (left ventricular ejection function (LVEF), left ventricular volumes, left ventricular regional wall motion, diastolic function (mitral inflow velocities as Early diastolic velocity (E), late diastolic velocity with atrial contraction (A), and deceleration time (DT), early diastolic velocity (e') and late diastolic velocity with atrial contraction (a') using tissue Doppler imaging, pulmonary artery systolic pressure (PASP), valvulopathy and aortic desease); assestment of risk stratification according to different scores (New York Heart Association (NYHA) classes, Canadian Cardiovascular Society (CCS) Angina grading scale, EUROSCORE II, American Society og Anesthesiologists (ASA) physical status classification system); preoperative patient therapy. In a following phase laboratory, hemodynamic and imaging evaluation will be carried out during and subsequent to CABG surgery. Through a coronary sinus inserted catheter will be dosed Troponine I (TnI) immediately before CPB and after the release of aortic cross clamp, about 10 minutes after the end of reperfusion. TnI will be also dosed at arrival on intensive care unit and 6, 12, 24, 48 h after unclamping of the aorta. Blood samples will be collected simultaneously from the radial artery and the coronary sinus before starting CPB and after removal of aortic cross clamp to evaluate lactates extraction, oxygen consumption (VO2) and oxygen extraction (O2ER), and C-reactive protein (CRP) pre and post-CPB. Hemodynamic measurements will be obtained by an arterial and a pulmonary artery catheter (PAC) inserted before surgery, and will include arterial pressure (systolic, diastolic and mean pressure), pulmonary artery pressure (PAP), right atrial pressure (RAP), pulmonary artery wedge pressure (PAWP), cardiac output (CO) and cardiac index (CI), systemic vascular resistance (SVR), left ventricular stroke work (LVSW), left stroke volume variaton (LSVV) and coronary artery perfusion pressure (CPP); these measurements will be conducted 30 min after intubation, after sternotomy, 10 min after protamin, after sternosynthesis, at arrival in the intensive care unit, 6, 12, 24, 36, 48 h after CPB. Lastly a transesophageal echocardiographic study will be performed by two expert echocardiographers following the protocols of the Society of Cardiovascular Anesthesiologists (21) and American Society of Echocardiography (22). Left ventricle myocardial performance index, LVEF, left ventricular regional wall motion, E/A ratio, E', E/E' and deceleration time (DT) of mitral inflow velocity will be measured; these measurements will be obteined 30 minute after intubation before sternotomy and ten minute after protamin. All collected data will be entered into a database in Excel format.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* sinus rhythm, heart rate (FC) ≥ 50 bpm at rest;
* NYHA class I, II, III (CCS I, II, III);

Exclusion Criteria:

* drugs intolerance or hypersensitivity;
* cardiogenic shock;ejection fraction (FE ) ≤ 50 % ;
* NYHA class IV (CCS IV);
* II or III atrioventricular block;
* a resting heart rate (HR) < 50 bpm or sick sinus syndrome;
* rate-corrected QT interval (QTc) greater than 500 ms;
* age <18 years;
* symptomatic hypotension or uncontrolled hypertension (systolic blood pressure at rest ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg);
* severe liver disease
* severe renal impairment (creatinine clearance ≤ 30 ml/min);
* from moderate to severe electrolyte disorders (potassium concentration < 2,5 or > 6 mmol/L; calcium concentration < 8 or > 11 mg/dl; magnesium < 1,8 or > 2,5 mg/dl);
* pregnancy;
* concomitant administration of potent CYP3A4 inhibitors (e.g. itraconazole, ketoconazole, voriconazole, posaconazole, HIV protease inhibitors, clarithromycin, telithromycin, nefazodone)
* concomitant administration of Class Ia (e.g. quinidine) or Class III (e.g. dofetilide, sotalol) antiarrhythmics other than amiodarone;
* previous cardiac interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Troponins I variation collected by coronary sinus pre and post clamping of the aorta. | Before cardiopulmonary by-pass and 10 minutes after the end of reperfusion
  A blood sample will be collected by coronary sinus and the sample sent by our laboratories to assess the concentration in µg/l of cardiac troponins directly in venous blood before cardiopulmonary by-pass and after the release of aortic cross clamp, about 10 minutes after the end of reperfusion.
Myocardial VO2 and O2 extraction variation collected by radial artery and coronary sinus pre and post clamping of the aorta. | Before cardiopulmonary by-pass and 10 minutes after the end of reperfusion
  Earlobe arterialized blood sample will be collected by radial artery coronary sinus and the sample sent by our laboratories to assess the concentration of VO2 and O2ER in ml/min in venous blood before cardiopulmonary by-pass and after the release of aortic cross clamp, about 10 minutes after the end of reperfusion.
Lactates variation collected by the radial artery and coronary sinus pre and post clamping of the aorta. | Before cardiopulmonary by-pass and 10 minutes after the end of reperfusion
  Earlobe arterialized blood sample will be collected by radial artery and coronary sinus and the sample sent by our laboratories to assess the concentration of lactates in mmol/L in venous blood before cardiopulmonary by-pass and after the release of aortic cross clamp, about 10 minutes after the end of reperfusion.
Troponins I variation collected by blood sample | Since arrival on intensive care unit and 6, 12, 24, 48 h after unclamping of the aorta
  A blood sample will be collected by peripheral vein and the sample sent by our laboratories to assess the concentration in µg/l of cardiac troponins Since arrival on intensive care unit and 6, 12, 24, 48 h after unclamping of the aorta.

SECONDARY OUTCOMES:
Echocardiographic evaluation to assess significant differences in terms of systolic and diastolic left ventricular function post cardiopulmonary by-pass. | 30 minute after intubation before sternotomy and ten minute after protamin
  Transesophageal echocardiographic study will be performed by two expert echocardiographers following the protocols of the Society of Cardiovascular Anesthesiologists and American Society of Echocardiography. Left ventricle myocardial performance index, LVEF (%), left ventricular regional wall motion, E/A ratio, E', E/E' and deceleration time (DT) of mitral inflow velocity will be measured; these measurements will be obteined.
Hemodynamic measurements | 30 min after intubation, after sternotomy, 10 min after protamin, after sternosynthesis, at arrival in the intensive care unit, 6, 12, 24, 36, 48 h after CPB
  Hemodynamic measurements will be obtained by an arterial and a pulmonary artery catheter (PAC) inserted before surgery, and will include arterial pressure (systolic, diastolic and mean pressure), pulmonary artery pressure (PAP), right atrial pressure (RAP), pulmonary artery wedge pressure (PAWP), cardiac output (CO) and cardiac index (CI), systemic vascular resistance (SVR), left ventricular stroke work (LVSW), left stroke volume variaton (LSVV) and coronary artery perfusion pressure (CPP).
Cardiac Complications | Since arrival on intensive care unit and 6, 12, 24, 48 h after unclamping of the aorta
  New-onset atrial fibrillation, ventricular arrhythmia, low cardiac output syndrome (LCOS), inotropic support and/or intraaortic balloon pump >24 hours, myocardial infarction) and intensive care unit and hospital length of stay between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Arlotta, MD, Study Director — Department cardiovascular diseases A. Gemelli Polyclinic , University Sacred Heart in Rome

IPD SHARING:
Plan to Share IPD: Yes